CLINICAL TRIAL: NCT01589536
Title: Improvement of the Social Medical Progression of Coronary Heart Disease With Associated Psychosocial Comorbidity by the Use of Interval Rehabilitation.
Brief Title: Social Medical Progression of Coronary Heart Disease With Associated Psychosocial Comorbidity -Interval Rehabilitation.
Acronym: SINKO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinic Roderbirken (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001
Record Dates: First submitted 2012-03-02; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Events
Keywords: psychocardiological; interval intervention; disability pension; risk profile; mental comorbidity
MeSH Terms: interventions — Comorbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventiongroup (Experimental): A Stationary psychocardiological interval-rehabilitation.
  Interventions: Other: interval-rehabilitation
- controlgroup (No Intervention): The Patients in the control group receive a personal recommendation concerning psychotherapy outpatient counseling and therapy services at home and take therapeutic help.

INTERVENTIONS:
Other: interval-rehabilitation — The Patients in the intervention group receive a Stationary psychocardiological interval-rehabilitation.The Interval rehabilitation is divided into individual psychological therapy with focus of Behavior therapy and relaxation therapy.
  Other Names: psychocardiological; interval rehabilitation; Roderbirken; comorbidity; sarah
  Arms: Interventiongroup

SUMMARY:
The purpose of the study is to verfiy the hypothesis if a short intensive psychocardiological interval-intervention, combined with a structured follow up, decreases the rate of disability retirements caused by psychosocial co-morbidity of patients with coronary heart disease.

DETAILED DESCRIPTION:
The purpose of the study is to verfiy the hypothesis if a short intensive psychocardiological interval intervention, combined with a structured follow up, decreases the rate of disability retirements caused by psychosocial co-morbidity of patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease
* Disease-related psychosocial morbidity
* not a disability retirements
* Insured with the German Rheinland pension (deutsche Rentenversicherung Rheinland)
* Sufficient language skills
* Age 18-58

Exclusion Criteria:

* Acute cardiac decompensation
* consuming the underlying disease
* psychotic disorder
* Acute suicidality
* pregnancy

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of the social medical progression of coronary heart disease with associated psychosocial comorbidity by the use of interval rehabilitaion | 24 months after including study
  Reducing the rate of disability pension of 18%of 9% by interval-rehabilitation with aftercare.

SECONDARY OUTCOMES:
Improvement of the social medical progression of coronary heart disease with associated psychosocial comorbidity by the use of interval rehabilitaion | 24 months after including study
  Reduction of cardiovascular events, including deaths Improving the risk profile Improvement of health-related quality of life Improvement of mental comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Mayer-Berger, MD, Principal Investigator — Clinic Roderbirken
Locations (1):
- Clinic Roderbirken, Leichlingen, North Rhine-Westphalia, Germany